CLINICAL TRIAL: NCT00000883
Title: Long-Term Assessment for Metabolic, Cardiovascular and Neurologic Complications In Subjects With Past CD4 Cells/mm3 Below 50 Who Increased CD4 Cells/mm3 to Above 100 on HAART
Brief Title: Long-Term Assessment for Metabolic, Cardiovascular and Neurologic Problems in HIV-Infected Patients With Increased CD4 Cells Counts Following Anti-HIV Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 362
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Antibiotics, Macrolide; Acquired Immunodeficiency Syndrome; Azithromycin; CD4 Lymphocyte Count; Anti-HIV Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
The purpose of this study is to see if there are any changes in sugar and fat levels in the blood when patients take anti-HIV therapy for many years. Another goal is to test memory and mental concentrations to determine if anti-HIV drugs protect the brain from damage caused by HIV.

(The purpose of this study has been changed from the original version.) HIV-infected patients with low CD4 cell counts are at risk for getting opportunistic (AIDS-related) infections. CD4 cells are cells of the immune system that help fight infection. Anti-HIV therapy may increase CD4 counts, which may lead to a decrease in AIDS-related infections. Problems that anti-HIV therapy is associated with include metabolic problems, neurologic problems, abnormal opportunistic infections, and cancer. Patients in ACTG 362 have been exposed to anti-HIV therapy longer than any other large group in the ACTG. These patients appear to benefit from their therapy, but also suffer problems from it. Observation of these patients should provide more information about long-term anti-HIV treatment and may detect unexpected problems.

(This study as been changed. More information about the reasons for conducting this study has been added.)

DETAILED DESCRIPTION:
The currently available data on clinical events in patients receiving potent antiretroviral therapy suggest that an alteration in the presentation of MAC disease may be seen and that rates of MAC disease may be reduced when patients respond to antiretroviral therapy. However, the extent of the protection and the timing of protection after initiation of therapy remain unknown. The current study should provide validated measures of immune restoration and clinical data to guide prophylaxis decisions for the many patients who are now responding to therapy after years of immune depletion. [AS PER AMENDMENT 11/16/99: The low rate of MAC in ACTG 362 patients after an average of 1 year of follow-up suggests that prophylaxis specifically for MAC disease with azithromycin is not necessary for patients who have experienced immune reconstitution. Prolonged follow-up will define durability of the antiretroviral response and the experience with opportunistic conditions, neurologic diseases, and survival, especially in those whose CD4 counts drop below 50 cells/mm3. It will also allow assessment of the levels of CD4 cell number at which vulnerability to opportunistic infection recur.] [AS PER AMENDMENT 03/18/03: During the extension of ACTG 362, serious complications of HAART have become better defined, including metabolic complications, neurologic problems, atypical opportunistic infections, and malignancies. Patients in ACTG 362 have been exposed to HAART longer than any other large group in the ACTG, and appear to benefit from and suffer complications of their therapy. Continued observation should provide estimates of expected complications and durability of long-term potent antiretroviral treatment, and may detect unanticipated problems.]

Patients are stratified at baseline for prior use of MAC into 3 groups: no prophylaxis, prior azithromycin prophylaxis, and other MAC prophylaxis. Patients are randomized to receive azithromycin (Arm I) or matching placebo (Arm II) once weekly and are followed every 8 weeks until study closure or for 18 months (72 weeks) after the last patient is enrolled. Patients who develop a drop in CD4 count below 50 cells/mm3 on 2 measurements at least 4 weeks apart are offered open-label azithromycin. [AS PER AMENDMENT 06/24/98: Patients remain on open-label azithromycin regardless of subsequent CD4 counts.] [AS PER AMENDMENT 11/16/99: The phase of Version 1.0 or Version 2.0 in which patients receive blinded-study medication is now referred to as Step I. The phase of Version 1.0 or Version 2.0 in which patients receive open-label azithromycin is now referred to as Step 2. Patients not currently on open-label azithromycin provided by the study enter Step 3 and discontinue study drugs, but remain blinded to the original treatment and are followed at 16-week intervals until study closure which will occur in April 2002 (3 years following enrollment of the last study participant). Any patient who develops a drop in CD4 count below 50 cells/mm3 on 2 measurements at least 4 weeks apart is offered open-label azithromycin. Patients currently receiving open-label azithromycin and patients from Step 3 who are initiating open-label azithromycin enter Step 4.] Patients undergo regular clinical and laboratory evaluations that include physical examinations, CD4 counts, and viral load. [AS PER AMENDMENT 11/16/99: Patients undergo clinical and laboratory evaluations every 16 weeks for 160 weeks that include physical examinations, CD4 counts, and viral load as well as neuropsychologic and cardiovascular assessments.] [AS PER AMENDMENT 01/18/01: All patients enrolled in the study are followed until April 2002.] [AS PER AMENDMENT 03/18/02: All patients currently participating in ACTG 362 are invited to continue follow up for an additional 5 years. Patients not currently receiving open-label azithromycin enter Step 5. Patients currently receiving open-label azithromycin enter Step 6, and continue to receive open-label treatment throughout the study. Any patient who enters on Step 5 and develops a drop in CD4 below 50 cells/mm3 on 2 consecutive measurements at least 4 weeks apart is offered open-label azithromycin and enters Step 6. Patients are assessed for metabolic, cardiovascular, and neurologic complications and are evaluated for opportunistic infections, CD4 counts, and viral load. Study visits occur at 32-week intervals until study closure.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 13 years old (need consent of parent or guardian if under 18).
* Have had an increase in CD4 cell count from less than or equal to 50 cells/mm3 to over 100 cells/mm3 on 2 separate occasions, at least 4 weeks apart. (This reflects a change in the CD4 cell count requirement.)
* Are on anti-HIV therapy.
* Are currently enrolled in Version 4.0 of the study.
* (This study has been changed to include the enrollment of patients into Version 4.0 of the study.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are allergic to azithromycin.
* Have had MAC disease.
* Have a history of tuberculosis (unless successfully treated and off anti-tuberculosis drugs for over 6 months) or other mycobacterial infection requiring chemotherapy.
* Have taken interleukin-2 (IL-2) in the past. (This study has been changed. Patients can now take IL-2 during the study.)
* Are taking certain medications.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 636
Dates: Start 1997-10; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Currier, Study Chair; Allen McCutchan, Study Chair; Susan Koletar, Study Chair
Locations (51):
- United States (51):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] von Reyn CF, Williams P, Becker S, Nevin T, Lederman H, Currier J. Skin test reactivity to mycobacterium avium sensitin among patients in ACTG 362. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:151 (abstract no 443)
- [Background] Cohn SE, Kammann E, Williams P, Chesney MA, Currier J. Predictors of adherence to azithromycin prophylaxis for prevention of mycobacterium avium complex (MAC) disease. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:151 (abstract no 444)
- [Background] Lederman HM, von Reyn CF, Becker S, Williams P, Currier J. Improved immunologic function correlates with CD4 rise after highly active anti-retroviral therapy (HAART). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:129 (abstract no 326)
- [Background] Currier JS, Williams PL, Koletar SL, Cohn SE, Murphy RL, Heald AE, Hafner R, Bassily EL, Lederman HM, Knirsch C, Benson CA, Valdez H, Aberg JA, McCutchan JA. Discontinuation of Mycobacterium avium complex prophylaxis in patients with antiretroviral therapy-induced increases in CD4+ cell count. A randomized, double-blind, placebo-controlled trial. AIDS Clinical Trials Group 362 Study Team. Ann Intern Med. 2000 Oct 3;133(7):493-503. doi: 10.7326/0003-4819-133-7-200010030-00008. PMID 11015162
- [Result] Cohn SE, Jiang H, McCutchan JA, Koletar SL, Murphy RL, Robertson KR, de St Maurice AM, Currier JS, Williams PL. Association of ongoing drug and alcohol use with non-adherence to antiretroviral therapy and higher risk of AIDS and death: results from ACTG 362. AIDS Care. 2011 Jun;23(6):775-85. doi: 10.1080/09540121.2010.525617. PMID 21293986